CLINICAL TRIAL: NCT04623320
Title: Validation of a 13C Glucose Breath Test to Quantify Insulin Resistance in Type 1 Diabetes Mellitus Compared With the Euglycaemic Clamp Test
Brief Title: Validation of a 13C Glucose Breath Test Compared With the Euglycaemic Clamp Test
Acronym: BRECLAIR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: 20/40/515
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-02

CONDITIONS: Insulin Resistance; Type 1 Diabetes
Keywords: insulin resistance; type 1 diabetes; euglycaemic clamp; breath test
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NAFLD+T1DM+: Subjects with type 1 diabetes and ultrasound-defined NAFLD
  Interventions: Diagnostic Test: euglycaemic clamp test; Diagnostic Test: 13C glucose breath test
- NAFLD-T1DM+: Subjects with type 1 diabetes without ultrasound-defined NAFLD
  Interventions: Diagnostic Test: euglycaemic clamp test; Diagnostic Test: 13C glucose breath test

INTERVENTIONS:
Diagnostic Test: euglycaemic clamp test — clamp test (golden standard) to determine insulin resistance
Diagnostic Test: 13C glucose breath test — 13C glucose breath test to compare with the golden standard

SUMMARY:
Insulin resistance can be assessed by the euglycaemic clamp technique. To date, this is the golden standard, but it is not suited for clinical practice. A 13C glucose breath test will be tested as a valid alternative. The curve of the exhaled 13C CO2 as a function of glucose metabolism can be correlated to the curve of the glucose disposal rate obtained via the clamp technique.

DETAILED DESCRIPTION:
The hyperinsulinemic-euglycemic clamp technique is the golden standard to assess insulin resistance in type 1 diabetes subjects. The plasma insulin concentration is acutely raised and maintained at 100 μU/ml by a continuous infusion of insulin. Meanwhile, the plasma glucose concentration is held constant at basal levels by a variable glucose infusion. When the steady-state is achieved, the glucose infusion rate equals glucose uptake by all the tissues in the body and is therefore a measure of tissue insulin sensitivity.

These data will be compared with the results of a 13C glucose breath test. Breath tests using 13C substrates are based on the principle that 13C CO2 in the exhaled breath can be measured as a metabolic tracer.

Breath testing has a major advantage over the clamp test in that it can be performed non-invasively and repeatedly without necessary supervision by medical staff.

ELIGIBILITY:
Inclusion Criteria:

* Adult type 1 diabetes patients
* 25/50 subjects with confirmed NAFLD (using ultrasound criteria)

Exclusion Criteria:

* pregnancy
* gastric bypass surgery
* cirrhosis
* secondary cause of liver steatosis present
* any cause which makes a 4-hour clamp impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 diabetes subjects from the research facility's outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of the 13C breath test with the golden standard | one day
  sensitivity and specificity analysis using linear regression

CONTACTS AND LOCATIONS:
Overall Officials: Christophe De Block, Prof., Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hussain M, Jangorbhani M, Schuette S, Considine RV, Chisholm RL, Mather KJ. [13C]glucose breath testing provides a noninvasive measure of insulin resistance: calibration analyses against clamp studies. Diabetes Technol Ther. 2014 Feb;16(2):102-12. doi: 10.1089/dia.2013.0151. Epub 2013 Oct 11. PMID 24116833
- [Background] Maldonado-Hernandez J, Martinez-Basila A, Salas-Fernandez A, Navarro-Betancourt JR, Pina-Aguero MI, Bernabe-Garcia M. The 13C-Glucose Breath Test for Insulin Resistance Assessment in Adolescents: Comparison with Fasting and Post-Glucose Stimulus Surrogate Markers of Insulin Resistance. J Clin Res Pediatr Endocrinol. 2016 Dec 1;8(4):419-424. doi: 10.4274/jcrpe.3260. Epub 2016 Jun 29. PMID 27354200
- [Result] Lewanczuk RZ, Paty BW, Toth EL. Comparison of the [13C]glucose breath test to the hyperinsulinemic-euglycemic clamp when determining insulin resistance. Diabetes Care. 2004 Feb;27(2):441-7. doi: 10.2337/diacare.27.2.441. PMID 14747226
- [Derived] Mertens J, Roosens L, Braspenning R, Vandebeeck J, Francque S, De Block C. The 13C Glucose Breath Test Accurately Identifies Insulin Resistance in People With Type 1 Diabetes. J Clin Endocrinol Metab. 2025 Jan 21;110(2):e432-e442. doi: 10.1210/clinem/dgae175. PMID 38487831
- [Derived] Clinck I, Mertens J, Wouters K, Dirinck E, De Block C. Insulin Resistance and CGM-Derived Parameters in People With Type 1 Diabetes: Are They Associated? J Clin Endocrinol Metab. 2024 Oct 15;109(11):e2131-e2140. doi: 10.1210/clinem/dgae015. PMID 38198792